CLINICAL TRIAL: NCT01722032
Title: Healthy Caregivers/Healthy Children
Brief Title: USDA Healthy Caregivers/Healthy Children: A Childhood Obesity Prevention Program
Acronym: HC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Stephanie Scott, Assistant Research Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009-05065
Record Dates: First submitted 2012-10-26; First posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Childhood Obesity
Keywords: childhood obesity, early childhood, nutrition
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The intervention centers' menus were modified to include more fresh fruit, fresh vegetables, low-fat (1%) or skim milk, water, less juice, and less simple carbohydrate snacks. The centers were also encouraged to incorporate fresh fruits and vegetables as often as possible for snack and meal time.
  Physical Activity. Physical activity was promoted for at least 60 minutes per day. TV viewing, watching movies and playing computer games were logged and limited to 30 minutes or less per day. Schools adopted "Best-Practice Policies".
  Interventions: Other: Childhood Obesity
- Control (No Intervention): Those schools randomized to the control arm received a safety curriculum and some child care center locations received an attention control consisting of three visits from the University of Miami Safety Van which provided parents and teachers with home, car and child seat safety information. The control group received all the same pre-post measures as the intervention arms. They also received the same incentives as the intervention arms to foster involvement and ensure retention/reduce loss to follow up.

INTERVENTIONS:
Other: Childhood Obesity
  Arms: Treatment

SUMMARY:
Background: Many unhealthy dietary and physical activity habits that foster the development of obesity are established by the age of five. Presently, approximately 70 percent of children in the United States are currently enrolled in early childcare facilities, making this an ideal setting to implement and evaluate childhood obesity prevention efforts. We describe here the methods for conducting an obesity prevention intervention randomized trial in the child care setting.

Methods/Design: A randomized, controlled obesity prevention trial in 28 low-income, ethnically diverse child care centers located throughout Miami-Dade County, FL is currently being conducted over two years (2010-present) to test the efficacy of an intervention that poises teachers and parents as lifestyle change agents. The Healthy Caregivers-Healthy Children (HC2) program includes a curriculum focusing specifically on healthy food choices, increased exercise, and role modeling. The program targets food policy changes throughout the school, and via the child, caregiver, and teacher. Major outcome measures include child body mass index percentile and z score, fruit and vegetable and other nutritious food intake, and amount of physical activity.

Discussion: Although few attempts have been made to prevent obesity during the first years of life, this period may represent the best opportunity for obesity prevention. Findings from this investigation should inform both the fields of childhood obesity prevention and early childhood research about the effects of an obesity prevention program housed in the childcare setting. (H1) A child care center-based obesity prevention intervention program that includes a teacher and parent nutritional gatekeeper and role modeling program will be more effective in maintaining BMI in 3-5 year olds compared to a control group.

(H2) Role modeling (teacher and parent) will be identified as a significant mediator in preventing obesity among intervention children versus controls.

(H3) A child care center-based multi-level obesity prevention intervention program will improve child nutrition (increased consumption of fruits and vegetables, decreased consumption of sweetened beverages) and increase physical activity level compared to a control group.

DETAILED DESCRIPTION:
Over one third of preschoolers were either overweight (18.4%) or obese (16.5%). The majority (92%) of caregivers of an overweight/obese child inaccurately perceived that their child was in a normal BMI category. Foreign-born caregivers were significantly more likely to inaccurately perceive their child's BMI percentile category, versus US-born caregivers (OR=0.65, 95% CI, 0.48-0.88). Specifically, those born in South America [OR=0.59. 95% CI, 0.36-0.98), Central America/Mexico (OR=0.59, 95% CI,0.41-0.85), and Caribbean Hispanic nations [OR=0.54, 95% CI 0.35-0.83) were significantly less likely to accurately perceive their child's BMI category, versus US-born caregivers.

Conclusions: The results of this study suggest that foreign-born parents of preschool-age overweight/obese children in particular do not accurately perceive their child's BMI status. Pediatricians and other healthcare providers serving foreign-born caregivers may consider additional healthy weight counseling for these families.

ELIGIBILITY:
Inclusion Criteria. Centers must have met the following criteria to be included: (1) have > 30 children ages 2-5 enrolled; (2) Serve low income families who are a part of the USDA food program and SNAP eligible; (3) Reflect the ethnic distribution of the Miami-Dade County Public School System (63 percent Hispanic, 19 percent African American, 18 percent white); and (4) Center directors agree to participate and sign a letter of commitment. Studies were excluded if they did not meet these criteria.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1100 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maintenance of a Child's Body Mass Index as a result of the intervention | up to two years
  Assessment of demographic variables, anthropometrics, food insecurity and parent perception were performed. Sociodemographic variables included age and gender of the children, country of birth of parent and child, years living in the US, and parental education (highest grade completed).
  Child Health Measures:Anthropometric Variables. Assessment of body composition included height (by stadiometer), weight (by digital scale), which was converted to BMI (weight in kilograms/height in meters squared) and then to a BMI age-and sex-adjusted BMI percentile. Participants were asked to remove shoes and any heavy outer clothing prior to measurement. Weight and height measurements were collected by trained staff based on US Department of Health and Human Services (HHS) guidelines for accurate anthropomorphic measurement. Research grade stadiometers and scales were used, and were brought from site to site by the staff.

SECONDARY OUTCOMES:
A Parent's perception of his/her child's weight status | up to two years
  Caregiver Measures. To assess parent perception of child weight status, the child's actual weight status (determined by BMI percentile group) was compared to the caregivers' response to the question "Do you consider your child to be overweight, underweight or about right weight for (his/her) age?" Food insecurity was measured by the short form of the USDA's Food Security Scale. This information was obtained by means of a structured parent interview or a self-administered survey. Caregiver BMI was obtained by self reported height and weight included on the caregivers survey. Parent acculturation was measured by items from the Stephenson Acculturation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Natale, PhD, Principal Investigator — University of Miami

REFERENCES:
- [Derived] Natale R, Scott SH, Messiah SE, Schrack MM, Uhlhorn SB, Delamater A. Design and methods for evaluating an early childhood obesity prevention program in the childcare center setting. BMC Public Health. 2013 Jan 28;13:78. doi: 10.1186/1471-2458-13-78. PMID 23356862